CLINICAL TRIAL: NCT04254549
Title: Evaluating the Therapeutic Efficacy of Rifaximin in Patients With Diabetic Gastroparesis Using Bloating as the Primary Endpoint.
Brief Title: Rifaximin in Patients With Diabetic Gastroparesis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor discontinued placebo. Unable to meet enrollment goals.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Lacy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-002908
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease; Diabetic Gastroparesis
MeSH Terms: conditions — Crohn Disease | interventions — Rifaximin; izencitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention Treatment (Experimental): Subjects diagnosed with gastroparesis will receive Rifaximin
  Interventions: Drug: Rifaximin
- Placebo Group (Placebo Comparator): Subjects diagnosed with gastroparesis will receive a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — 550 mg by mouth three times daily for 14 days
  Other Names: TD-1473
  Arms: Intervention Treatment
Drug: Placebo — By mouth three times daily for 14 days
  Arms: Placebo Group

SUMMARY:
Researchers are trying to determine if subjects with diabetic gastroparesis and symptoms of bloating will have a greater improvement in bloating symptoms when treated with rifaximin.

ELIGIBILITY:
Inclusion Criteria

* Men and women adult patients, aged 18-75, with diabetic gastroparesis
* Diagnosis of diabetic gastroparesis will have been made previously using a combination of symptoms (e.g., nausea, vomiting, bloating, early satiety, abdominal pain), the absence of mechanical obstruction, and delayed gastric emptying using a 4-hour, solid phase scintigraphic study (GES; > 20% remaining at 4 hours)

Exclusion Criteria

* Prior surgery to the stomach or esophagus
* Known mechanical obstruction of the GI tract
* Current or recent (< 4 weeks) use of opioids
* Current/active use of cannabis
* Current or recent (< 4 weeks) use of antibiotics
* Current or recent use of antifungal agents (< 4 weeks)
* Prior treatment with rifaximin (< 1 year)
* Uncontrolled diabetes with a HgbA1c > 12
* Severe uncontrolled or untreated anxiety or depression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Improvement in bloating | Week 2, week 4, week 8
  Change is the self reported bloating questionnaire comprised of 45 questions addressing symptoms of bloating/distention

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Lacy, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials